CLINICAL TRIAL: NCT06292338
Title: A Comparative Study of Lung Ultrasound in Assessment of Neonatal Respiratory Disorders With Other Diagnostic Aids in NICU of Assuit University Children's Hospital
Brief Title: Lung Sonar in Neonatal Respiratory Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Gehad Adel Mohammed Hussein (Other)
Responsible Party: Sponsor-Investigator, Gehad Adel Mohammed Hussein, Specialist of pediatrics, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AUCHAU
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Respiratory Distress
Keywords: LUS; Neonates; Respiratory disorders
MeSH Terms: conditions — Pulmonary Atelectasis; Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to determine the value of chest ultrasonography in comparison to other tools as chest x-ray and ABG in diagnosis and follow up of neonates with respiratory disorders.

DETAILED DESCRIPTION:
Respiratory distress is the most frequent cause of neonatal intensive care unit (NICU) admission, and the individual management strategies should be the main task in NICUs for these infants. Fifteen percent of term infants and twenty-nine percent of late preterm infants admitted to the NICU develop significant respiratory morbidity; this is even higher for infants born before 34 weeks' gestation. Neonatal respiratory distress syndrome (NRDS) is one of the most common causes of neonatal respiratory failure and neonatal mortality, especially in premature infants, who tend to have very low birth weight.NRDS is a pulmonary insufficiency caused by structural and functional immaturity of the lung. The incidence of NRDS depends upon gestational age and varies from 92% for infants born at 24-25 weeks to 57% for those born at 30-31 weeks.Mortality from NRDS varies according to the infants' weight, from 50% for infants of <1.0 kg to 0% for those of more than 4.0 kg.Infants affected by NRDS usually require pulmonary surfactant and continuous positive airway pressure (invasive ventilation or mechanical ventilation). Although chest X-Ray plays an important role in diagnosis of respiratory distressed neonates, it leads to their exposure to ionizing radiation due to their small size and the close proximity of radiosensitive tissues and organs are at greater risk from latent effects of chest Xray in comparison to other age groups. As chest x-ray (CXR) and/or chest computerized tomography (chest CT) are the main imaging tools in the diagnosis of lung diseases. For a long time, the lung ultrasound (LUS) was considered a "forbidden zone" in the diagnosis of lung diseases since ultrasonic waves are totally reflected when encountering air. However, by utilizing ultrasonic artefacts formed by different pathological changes in adults, children and poor newborn infants,this "forbidden zone" has been contested and point-of-care lung ultrasound (POC-LUS) has been successfully used for the diagnosis of lung diseases. Neonatal lung ultrasound (LUS) is used in emergent situations, differentiating neonatal respiratory pathologies, and predicting neonatal morbidity . LUS can be brought to the bedside of the fragile neonate, used serially, and does not expose the neonate to ionizing radiation.

Functional and descriptive applications make it a high-fidelity tool to aid in distinguishing the various causes of neonatal respiratory failure and to guide in management . LUS also has increased sensitivity and specificity in comparison with an X-ray for the detection of respiratory pathologies (e.g., TTN , RDS, pmeumothorax, and pleural effusion) and can be utilized to monitor progress of clinical pathologies.The neonatologist-performed LUS has the advantage of being immediately interpreted by those caring for the neonate, potentially leading to more accurate diagnosis and timely therapeutic as intervention. One of the most important applications is the recently proposed use of the LUS score as a semiquantitative assessment of the severity of lung diseases. Efforts have been made to determine the relationship between these scores and the diagnosis of the disease . This study aimed to evaluate the relationship between the LUS score and the diagnosis of neonates hospitalized because of respiratory disorder.

In this study, the investigators also aimed to evaluate the correlation between LUS scores and blood gas parameters in patients hospitalized for respiratory distress and to get an idea about the severity of the disease.Therefore, it can be used to predict the need for surfactants in preterm infants. Its positive role in predicting surfactant need in very- and extremely preterm newborns disease and also the development of chronic lung disease in preterm neonates has been reported recently . LUS scores obtained during the first days of life can provide information about the prognosis of neonatal respiratory failure and predict the need for respiratory support . In addition, LUS performs a useful role in predicting non-invasive ventilation failure in neonates with respiratory distress, and this is important for the clinician to decide to apply invasive mechanical ventilation to prevent clinical deterioration . Lung ultrasound has a prognostic value in monitoring and follow-up of lung development in preterm infants. and it is an adequate tool to predict the development of bronchopulmonary dysplasia (BPD)in infants born preterm before 32 weeks of gestation: for diagnosis of BPD from as early as 3 days post birth, although the optimal timing for its use is 1 week post birth .

The usual evolution of pulmonary patterns in neonates delivered before 32 weeks starts with a pattern characteristic of RDS at birth, with high LUS score values in the 1st days, but then normally improve thereafter as the primary surfactant deciency resolves, reaching LUS score values near 0 at around 1 week post birth.The patients whose LUS scores do not exhibit this decrease or actually increase are more likely to develop BPD.

ELIGIBILITY:
Inclusion Criteria:

* neonates with a gestational age ≥28 weeks who are suffering from respiratory disorders.

Exclusion Criteria:

* neonates having multiple congenital anomalies, chromosomal aberrations, hydrops fetalis and/or heart failure.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates (Term and preterm) presented with respiratory disorders
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparing between LUS and Chest xRay in neonatal respiratory disorders assessment | 1 year
  Our study aimed to evaluate the relationship between the LUS score and the diagnosis of neonates hospitalized because of respiratory disorder.
  In our study, we also aimed to evaluate the correlation between LUS scores and blood gas parameters in patients hospitalized for respiratory distress and to get an idea about the severity of the disease.